CLINICAL TRIAL: NCT07379190
Title: Efficacy and Safety of Tirofiban Therapy in Acute Ischemic Stroke Patients Beyond the Time Window Guided by High-Resolution Magnetic Resonance Imaging
Brief Title: HR-MRI-Directed Tirofiban Therapy for Late-Window Acute Ischemic Stroke (TIAN)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weifang Medical University (Other)
Collaborators: Linyi People's Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Weili Li, Professor, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TITAN
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Cerebral Infarction
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebral Infarction | interventions — Tirofiban; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban Combined with Standard Medication Therapy Group (Experimental): Patients were randomized to the Tirofiban Combined with Dual Antiplatelet Therapy Group. Intravenous tirofiban was administered within 30 minutes of randomization, with an initial bolus infusion at a rate of 0.4 μg/(kg·min) for 30 minutes, followed by a continuous infusion at 0.1 μg/(kg·min) for 47.5 hours. During this period, dual antiplatelet therapy (DAPT) was initiated at a dose of aspirin 100 mg/day plus clopidogrel 75 mg/day, with an overlapping duration of 4-6 hours. After the completion of tirofiban infusion, dual antiplatelet therapy (aspirin 100 mg/day plus clopidogrel 75 mg/day) was continued for a total of 21 days, followed by long-term maintenance with aspirin 100 mg/day alone.
  Interventions: Drug: Tirofiban; Drug: dual antiplatelet therapy
- Standard Medication Therapy Group (Active Comparator): Patients were randomized to the control group, with dual antiplatelet therapy (DAPT) initiated as early as possible at a dose of aspirin 100 mg/day plus clopidogrel 75 mg/day for a total of 21 days, followed by long-term maintenance with aspirin 100 mg/day alone.
  Interventions: Drug: dual antiplatelet therapy

INTERVENTIONS:
Drug: Tirofiban — Intravenous tirofiban was administered within 30 minutes of randomization, with an initial bolus infusion at a rate of 0.4 μg/(kg·min) for 30 minutes, followed by a continuous infusion at 0.1 μg/(kg·min) for 47.5 hours.
  Arms: Tirofiban Combined with Standard Medication Therapy Group
Drug: dual antiplatelet therapy — Initiate dual antiplatelet therapy as early as possible (aspirin 100 mg/day plus clopidogrel 75 mg/day) for a total of 21 days, followed by long-term maintenance with aspirin 100 mg/day alone. For patients at high risk of stroke, such as those with severe stenosis of major blood vessels, dual antiplatelet therapy should be administered for 90 days.
  Other Names: aspirin; clopidogrel

SUMMARY:
This study aims to address the existing clinical challenges by introducing high-resolution magnetic resonance vessel wall imaging (HR-MRI), an advanced imaging technology, to achieve precise etiological classification in patients with acute ischemic stroke (AIS) beyond the time window. HR-MRI allows clear visualization of intracranial arterial wall structures and direct identification of key pathological features of the culprit vessel, including atherosclerotic plaques, vascular wall remodeling, and intracranial hemorrhage, thereby enabling reliable differentiation between intracranial atherosclerotic large artery atherosclerosis (ICAS-LAA) stroke and other etiological subtypes such as cardiogenic embolism. Based on the latest clinical demands and advances in imaging technology, this study intends to evaluate the efficacy and safety of tirofiban in patients with ICAS-LAA stroke beyond the time window under the precise guidance of HR-MRI. It is expected to provide high-level evidence-based medical evidence for this specific patient population and further optimize clinical diagnosis and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Acute ischemic stroke (AIS) in the anterior intracranial circulation (internal carotid artery system) confirmed by clinical symptoms and imaging examinations;
3. Time from symptom onset or last known normal state to randomization: > 24 hours and ≤ 7 days;
4. Stroke subtype confirmed as intracranial large artery atherosclerosis (ICAS) by high-resolution vessel wall imaging (HR-VWI) according to the TOAST classification, with cardiogenic embolism and other etiologies excluded;
5. Baseline National Institutes of Health Stroke Scale (NIHSS) score of 4-20 at the time of randomization;
6. Signed informed consent form obtained from the patient or their legal representative.

Exclusion Criteria:

1. Planned to receive reperfusion therapy (endovascular therapy or intravenous thrombolysis)；
2. Intracranial hemorrhage confirmed by computed tomography (CT)；
3. Definite or suspected cardiogenic embolism；
4. History of atrial fibrillation or current electrocardiogram indicating atrial fibrillation；
5. Acute ischemic stroke caused by other etiologies, such as Moyamoya disease, arterial dissection, arteritis, etc；
6. Imaging examinations indicating that the area of the current cerebral infarction exceeds 1/2 of the area of a single cerebral lobe;
7. Known contraindications to antiplatelet therapy, including hematochezia, gastrointestinal bleeding, or any other hemorrhagic disorders;
8. History of hypersensitivity to aspirin;
9. Definite indication for anticoagulant therapy expected during the study period (e.g., atrial fibrillation, mechanical heart valve, deep vein thrombosis, pulmonary embolism, antiphospholipid antibody syndrome, hypercoagulable state, etc.);
10. Complicated with malignant tumors, chronic hemodialysis, severe renal insufficiency (glomerular filtration rate [GFR] < 30 ml/min or serum creatinine [Cr] > 220 μmol/L (2.5 mg/dl)), or severe hepatic insufficiency (serum alanine aminotransferase [ALT] > 2 times the upper limit of normal [ULN], or serum aspartate aminotransferase [AST] > 2 times the ULN);
11. Severe heart failure (New York Heart Association [NYHA] Functional Classification Class III or IV);
12. Complicated with severe non-cardiovascular comorbidities, with an estimated survival time < 6 months;
13. Concurrent new cerebral infarction in both anterior and posterior circulations;
14. Inability to complete the follow-up procedures;
15. Presence of other known neurological disorders that may complicate the follow-up;
16. Concurrent participation in other therapeutic clinical trials with incomplete treatment and follow-up;
17. Other conditions that the investigators consider inappropriate for enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with functional independence outcome [modified Rankin Scale(mRS) score 0-1] | 90 ± 7 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death); a lower score indicates a better prognosis.

SECONDARY OUTCOMES:
Proportion of participants with good prognosis (mRS score 0-2) | 90 ± 7 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death);a lower score indicates a better prognosis.
Proportion of participants with mRS score 0-3 | 90 ± 7 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death);a lower score indicates a better prognosis.
Distribution of mRS scores | 90 ± 7 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability,and 6=death);a lower score indicates a better prognosis.
EuroQol Five-Dimension Questionnaire (EQ-5D) score | 90 ± 7 days after randomization
  The EQ-5D is a standardized patient-reported outcome measure for evaluating health-related quality of life (HRQoL), consisting of the EQ-5D descriptive system (assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and the EQ visual analog scale (EQ-VAS). The utility score derived from the descriptive system will be adopted for statistical analysis, with a range of -0.594 to 1.0 based on the applicable value set. A higher score indicates better health-related quality of life: a score of 1.0 represents perfect health, 0 equates to a health state equivalent to death, and negative scores reflect health states worse than death. The EQ-VAS (0-100 scale, 0 = worst imaginable health state; 100 = best imaginable health state) will be analyzed as a supplementary index.
Barthel Index (BI) score | 90 ± 7 days after randomization
  the BI is an ordinal disability score of 10 categories(range from 0 to 100, higher values indicate better prognosis);
Proportion of participants with neurological improvement within 24 hours of randomization [≥2-point reduction in National Institutes of Health Stroke Scale (NIHSS) score from baseline] | 24 ± 6 hours
  the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits);
National Institutes of Health Stroke Scale (NIHSS) scores | Time Frame: 24h; before discharge; day7
  NIHSS score increased by more than 4 points);the NIHSS is a stroke severity score composed of 11 items (range from 0 to 42, higher values indicate more severe deficits)
Proportion of participants with symptomatic intracranial hemorrhage (sICH) within 24 hours of randomization | 24 ± 6 hours
  clinical safety endpoint
Early neurological deterioration(END) | 24 ± 6 hours
  defined as NIHSS score increased by #4 points within 24 hours
Incidence of serious adverse events (SAEs) | 24 ± 6 hours;
  clinical safety endpoint
Incidence of any adverse events | 24 ± 6 hours;
  clinical safety endpoint
Recurrent stroke | 90 ± 7 days after randomization
  clinical safety endpoint;the new neurological deficit must be accompanied by corresponding new ischemic or hemorrhagic lesions on brain CT or MRI, which are not contiguous with the index stroke lesion and do not correspond to the vascular territory of the index stroke.
all-cause mortality; | 90 ± 7 days after randomization
  clinical safety endpoint; to observe the proportion of all patients who died in each group
stroke-related mortality | 90 ± 7 days after randomization
  clinical safety endpoint;The proportion of stroke related deaths in each group
Proportion of participants with any intracranial hemorrhage | 24 ± 6 hours
  imaging safety endpoints; to observe the proportion of intracranial hemorrhage patients in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Weifang People's Hospital, Weifang, China/Shandong Province, China